CLINICAL TRIAL: NCT05228275
Title: Prospective Cohort Study to Evaluate Immunologic Response Following COVID-19 Vaccination in Children, Adolescents and Young Adults With Cancer
Brief Title: Evaluation of Immunologic Response Following COVID-19 Vaccination in Children, Adolescents, and Young Adults With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCL21C2; NCI-2022-01919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL21C2 (Other: Children's Oncology Group); COG-ACCL21C2 (Other: DCP); ACCL21C2 (Other: CTEP); U24CA196173 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19 | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (survey, biospecimen collection): Patients receive COVID-19 vaccine per standard of care. Patients also complete a survey at 1 month and undergo collection of blood samples at 1, 3, 6, 12, 18, and 24 months. Patients may complete an additional survey at 1 month after each vaccine boost and undergo collection of blood samples before each vaccine boost, 1 month after each vaccine boost, and at the time of COVID-19 infection.
  Interventions: Procedure: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Survey Administration — Complete survey

SUMMARY:
This study evaluates immunologic response following COVID-19 vaccination in children, adolescents, and young adults with cancer. Vaccines work by stimulating the body's immune cells to respond against a specific disease. The immune response produces protection from that disease. Effects from cancer and from treatments for cancer can reduce the body's natural disease fighting ability (called immunity). Factors such as vaccine type, timing of vaccine dosing related to treatment for cancer and number of vaccine doses or "boosts" (extra vaccine shots) may strengthen or diminish the body's protective immune response. This study may help researchers learn more about how the body's immune system responds to the COVID-19 vaccine when the vaccination is given during or after cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize the immunologic response following severe acute respiratory syndrome (SARS)-coronavirus (CoV)-2 vaccination in children, adolescents, and young adults with cancer who are currently receiving or who recently completed treatment with immunosuppressive therapy.

EXPLORATORY OBJECTIVES:

I. Describe the rate of post-vaccination symptomatic SARS-CoV-2 infections. II. Assess the durability of immune response to SARS-CoV-2 vaccine over 2 years.

III. Describe the longer-term impacts of vaccine immune response including subsequent COVID-19-related serious illness.

IV. To help guide future vaccine dosing and timing, at each SARS-CoV-2 vaccine dose administration determine the degree of:

IVa. Lymphopenia (absolute lymphocyte count cells/mm^3); IVb. Helper T-cell suppression (CD4 count); IVc. B-cell suppression (CD19 count). V. Provide a mechanism for data collection and banking of biospecimens for use in research regarding immune response to SARS-CoV-2 vaccination.

OUTLINE:

Patients receive COVID-19 vaccine per standard of care. Patients also complete a survey at 1 month and undergo collection of blood samples at 1, 3, 6, 12, 18, and 24 months. Patients may complete an additional survey at 1 month after each vaccine boost and undergo collection of blood samples before each vaccine boost, 1 month after each vaccine boost, and at the time of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* >= 6 months and =< 37 years of age at time of enrollment
* Patient plans to receive their first COVID-19 vaccine dose one of the food and drug administration (FDA) approved/FDA-emergency use authorization (EUA) approved COVID-19 vaccines OR patient already received their first COVID-19 vaccine dose =< 24 months prior to enrollment using one of the FDA approved/FDA-EUA approved COVID-19 vaccines.

  * Note: for this observational study, the decision to vaccinate is according to local discretion and should be made prior to consideration of enrollment
* Must have a diagnosis of cancer
* Patient must be undergoing or have previously received one of the following cancer treatments within 12 months before their first COVID-19 vaccine dose:

  * Dosing with chemotherapy or immunotherapy agent, including tyrosine kinase inhibitors and small molecule inhibitors targeting cancer
  * Dosing with monoclonal antibodies targeting B-cell antigens (e.g., Rituximab), or Bruton tyrosine kinase inhibitors or Janus Kinase inhibitors
  * Stem cell infusion for bone marrow transplant or CAR-T infusion for cellular therapy
* A patient enrolling prior to their first COVID-19 vaccine dose is eligible only if it is feasible to collect required baseline study specimens within protocol mandated time period prior to the initial COVID-19 vaccine dose; or a patient who already received a COVID-19 vaccine is eligible only if feasible to collect at least one post-first-dose follow-up specimen (i.e., at minimum, collection of the 24m PFD follow-up specimen must be feasible as per timing requirements

  * Note: for this observational study, the vaccine timing and regimen will proceed according to local discretion. Patients enrolled prior to their first COVID-19 vaccine dose who do not receive initial vaccine dose within 3 months after enrollment will be taken off study
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, FDA, and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Documented SARS-CoV-2 monoclonal antibody infusion or convalescent plasma after COVID-19 infection within last 90 days

  * Note: patients with previous COVID-19 infection are eligible as long as requirements are met. Patients receiving intravenous immunoglobulin therapy (IVIG) therapy (i.e., post bone marrow transplantation [BMT] or chimeric antigen receptor [CAR]-T) are eligible
* Patients undergoing radiation therapy only are ineligible

  * Reminder: before the planned initial COVID-19 vaccine dose, patient must be undergoing or have received cancer treatments

Ages: 6 Months to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults with cancer receiving approved COVID-19 vaccines
Sampling Method: Non-Probability Sample
Enrollment: 549 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2-specific protective antibodies | 24 months following initial vaccination with a protocol-approved COVID-19 vaccine
  Will report the proportion of patients with a serologic response to a protocol-approved COVID-19 vaccine, captured using a test for SARS-CoV-2-specific antibodies via immunoassay, and will report a corresponding 95% confidence interval.

OTHER OUTCOMES:
Durability of immune response at 6 months | At 6, 12 and 18 months after each dose
  The proportion of patients with an immune response (seropositivity) at 6, 12 and 18 months after the initial dose will be calculated along with a corresponding 95% confidence interval.
Post-vaccination symptomatic SARS-CoV-2 infections | Up to 2 years after initial dose
  The proportion of patients with a post-vaccination symptomatic SARS-CoV-2 infection will be calculated along with a corresponding 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Emad K Salman, Principal Investigator — Children's Oncology Group
Locations (72):
- United States (72):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Illinois, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin